CLINICAL TRIAL: NCT03005639
Title: Neoadjuvant Vemurafenib and Cobimetinib in BRAF V600 Mutant Stage IIIB-C Melanoma
Brief Title: ML29255 Neoadjuvant Vemurafenib and Cobimetinib Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor has decided to close study.
Sponsor: Inova Health Care Services (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-2316
Record Dates: First submitted 2016-05-02; First posted 2016-12-29 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Stage IIIB-C Melanoma
MeSH Terms: interventions — Vemurafenib; cobimetinib

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vemurafenib/Cobimetinib (Experimental): Vemurafenib and cobimetinib as a combination has been approved by the United States Food and Drug Administration (FDA) for patients with more advanced melanoma. In this trial, vemurafenib and cobimetinib combination is considered to be experimental since safety of this combination prior to lymph node surgery has not been studied.
  Interventions: Drug: Vemurafenib and Cobimetinib

INTERVENTIONS:
Drug: Vemurafenib and Cobimetinib — All participants will receive study treatment for up to 56 days (8 weeks). After completing treatment, they will undergo a lymph node removal surgery. After surgery, they will have follow-up visit 2-4 weeks after surgery.
  Other Names: Zelboraf for vemurafenib

SUMMARY:
Neoadjuvant Vemurafenib and Cobimetinib in BRAF V600 Mutant Stage IIIB-C Melanoma

• To evaluate the overall radiological complete response rate in patients with stage IIIB/C melanoma after 8 weeks of neoadjuvant vemurafenib and cobimetinib

DETAILED DESCRIPTION:
Vemurafenib and cobimetinib are FDA-approved drugs to treat advanced melanoma that has a mutated (changed) form of a cell protein called BRAF (BRAF V600 mutation). The purpose of this study is to determine if vemurafenib and cobimetinib can be safely given to patients with this type of melanoma to shrink it before surgery. This research is being done because patients with melanoma spread to lymph node have high chance of melanoma recurrence even after lymph node removal surgery, and currently there is no approved medicine to use for patients with BRAF V600 mutant melanoma before lymph node removal surgery.

Vemurafenib and cobimetinib as a combination has been approved by the United States Food and Drug Administration (FDA) for patients with more advanced melanoma. In this trial, vemurafenib and cobimetinib combination is considered to be experimental since safety of this combination prior to lymph node surgery has not been studied.

Before the participant begins the study:

The participant will need to have the following exams, tests or procedures to find out if eligibility is met.

* A skin exam
* An eye exam
* An electrocardiogram (ECG) which is a test that tracks the electricity of the heart
* An echocardiogram (a test that uses sound waves to create pictures of the heart) or MUGA scan (a test that uses radioactive materials called tracers to show the heart chambers) which is a test to evaluate the function of the heart
* A blood test
* A biopsy of lymph node

If the exams and tests listed above show that the individual can take part in the study, and he or she chooses to take part, then the participant will take the study drugs for 8weeks. He/she will take vemurafenib 240mg 4tablets twice daily for 56days and cobimetinib 20mg 3 tablets daily on days 1-21 and 29-49. While taking these pills, the following extra exams and tests will be needed.

* Four extra blood samples will be drawn. One blood sample will be drawn immediately before the first dose of the vemurafenib and trametinib pills. Then blood sample will be drawn 2 weeks, 4weeks, and 8weeks after starting the pills.
* A biopsy of lymph node will be performed 2weeks after starting the pills.
* Skin exams will be performed immediately before the first dose, 2weeks, 4weeks, and 8weeks after starting the pills.
* Eye exams will be performed 4weeks, 8weeks after starting the pills.
* An ECG will be performed 2weeks, 4weeks, and 8weeks after starting the pills.
* An echocardiogram or MUGA scan will be performed 4weeks after starting the pills.
* A CT scan will be performed 8weeks after starting the pills.

Once the participant finishes 8weeks of study drugs, he or she will undergo surgery within a week. After surgery, the individual will need the following extra exam.

• A skin exam A blood sample will be taken for the study at the first study visit, two week visit and eight week visit. Tissue from a core biopsy will be taken for the study at the first study visit and two week visit. This sample is required in order for the individual to take part in this study because the research on the sample is an important part of the study. The research biopsy is done in a similar way to biopsies done for diagnosis. Neither the participant nor the participant's health care plan/insurance carrier will be billed for the collection of the blood and tissue sample that will be used for this study. The results will not be made available to the participant during participation in the trial.

ELIGIBILITY:
Patients will be included in the study based on the following criteria:

* Signed informed consent
* Histologically confirmed, palpable, regional lymph node metastatic melanoma ≥ 1.5cm (stage IIIB-C; N1b-3) either at initial presentation or at regional lymph node recurrence considered surgically resectable at baseline by the treating medical oncologist and surgical oncologist
* Patients with intransit or satellite metastases with lymph node involvement are allowed if considered surgically resectable at baseline
* Measurable disease per RECIST 1.1
* Melanoma must be documented to contain a BRAFV600 mutation by a CLIA approved laboratory
* No evidence of distant metastasis
* Age ≥ 18 years
* ECOG performance status ≤1
* Adequate bone marrow function as indicated by the following:

  * ANC greater than 1500/µL
  * Platelets ≥ 100,000/µL
  * Hemoglobin greater than 9 g/dL
* Adequate renal function, as indicated by creatinine ≤1.5 x the upper limit of normal (ULN)
* Adequate liver function, as indicated by bilirubin ≤1.5 x ULN
* AST or ALT less than 3 x ULN (patients with documented liver metastases: AST and/or ALT ≤5 x ULN)
* Able to swallow pills
* Negative serum pregnancy test within 7 days prior to commencement of dosing in premenopausal women. Women of non-childbearing potential may be included without serum pregnancy test if they are either surgically sterile or have been postmenopausal for ≥ 1 year.
* Fertile men and women must use an effective method of contraception during treatment and for at least 6 months after completion of treatment as directed by their physician. Effective methods of contraception are defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly (for example implants, injectables, combined oral contraception or intra-uterine devices). At the discretion of the Investigator, acceptable methods of contraception may include total abstinence in cases where the lifestyle of the patient ensures compliance. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Willing and able to undergo biopsy for research purposes
* Willing and able to sign informed consent

Exclusion Criteria:

* Had prior radiotherapy at lymph node basin
* Prior treatment with BRAF inhibitor or MEK inhibitor
* Active infection
* Pregnant, lactating or breast feeding women
* Concomitant malignancies or previous malignancies within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* History of malabsorption or other condition that would interfere with absorption of vemurafenib or cobimetinib
* Any underlying medical or psychiatric condition, which in the opinion of the Investigator will make the administration of vemurafenib and cobimetinib hazardous
* Unwillingness or inability to comply with study and follow-up procedures.
* The following foods/supplements are prohibited at least 7 days prior to initiation of and during study treatment:

  * St. John's wort or hyperforin (potent cytochrome P450 CYP3A4 enzyme inducer)
  * Grapefruit juice (potent cytochrome P450 CYP3A4 enzyme inhibitor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-02-24 (Actual); Study Completion 2018-02-24 (Actual)

PRIMARY OUTCOMES:
Radiologic Complete Response Rate | Day 56 (+/- 3 days)
  Radiologic complete response rate will be the primary endpoint. This will be assessed after completion of the 8-week treatment of vemurafenib and cobimetinib by CT measurements of tumor diameter pre-treatment and at day 56 (± 3 days) using RECIST 1.1. Complete response (CR) is defined by a reduction in the short-axis diameter of any pathologic lymph node to less than 10 mm, whereas partial response (PR) is defined as 30% or more decrease in the short axis. The analysis of response rate is based on the efficacy evaluable patients who has post-treatment CT scan at Day 43. Patients who discontinued study drug or withdraw from the study will be included only if they had post-treatment CT scan. We will calculate radiologic complete response rate with 95% confidence interval.

SECONDARY OUTCOMES:
Overall response rate, pathologic complete response rate | Day 56 (+/- 3 days)
  Overall response rate is defined as the proportion of the patients in the analysis population who have a CR or PR. Pathologic complete response is defined as the absence of any residual invasive cancer on hematoxylin and eosin evaluation of all sampled lymph nodes +/- primary melanoma specimen following completion of neoadjuvant systemic therapy (ypT0ypN0 in the current AJCC staging system). The analysis of pathologic response is based on the efficacy evaluable patients who underwent therapeutic lymph node dissection. Patients who discontinued study drug or withdraw from the study will be included only if they underwent therapeutic lymph node dissection. We will calculate the pathological complete response rate with 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Sekwon Jang, MD, Principal Investigator — Inova Schar Cancer Institute
Locations (1):
- Inova Schar Cancer Institute, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No